CLINICAL TRIAL: NCT05962411
Title: A Large-Scale Randomized Control Trial to Determine the Effects of Dress by Adolescents on Electronic Cigarette Retailer Behaviors in Regulation Compliance in China
Brief Title: Effects of Dress by Adolescents on Electronic Cigarette Retailer Behaviors in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: China Medical Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-430
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2023-07

CONDITIONS: Regulation Compliance; Electronic Nicotine Delivery Systems
Keywords: Electronic Cigarette; Retailer; Adolescent; Regulation Compliance; China
MeSH Terms: conditions — Vaping | interventions — Bandages

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dress in School Uniforms (No Intervention): Simulated clients dress in school uniforms, enter e-cigarette stores, and act as minor buyers.
- Dress in Professional Attire (Experimental): Simulated clients dress in business casuals, enter e-cigarette stores, and act as potential "adult e-cigarette buyers".
  Interventions: Other: Dress in Professional Attire

INTERVENTIONS:
Other: Dress in Professional Attire — "Adolescents" pretend to be "adult e-cigarette buyers" by dressing in professional attire.
  Arms: Dress in Professional Attire

SUMMARY:
This study is a national-level randomized control trial to measure the effects of dressing in professional attire by adolescents on regulation compliance-related behaviors of electronic cigarette (e-cigarette) retailers defined by both age verification and potential underage sales. The corresponding null hypothesis that will be tested is that dressing in professional attire by adolescents will have no effect upon retailer behaviors in regulation compliance. The secondary objectives are to determine the impacts of type of dress by adolescents on marketing and communication strategies adopted by retailers, as well as to document the differences in the behaviors between e-cigarette and tobacco retailers.

DETAILED DESCRIPTION:
Electronic cigarette (e-cigarette) use has been growing dramatically and poses a significant public health threat to adolescents in China. After the online sales of these products has been banned, purchases from brick-and-mortar stores became the only legal option for the users. However, little research has been conducted to document sales behaviors of the physical retailers and identify the associated factors. The study will investigate the extent to which dressing in professional attire by adolescents on regulation compliance in retailer behaviors, including inquiring about age, requesting identity cards for age verification, and completing transactions even when identity cards are not presented. Adopting the simulated client method, the study will collect information on regulation compliance, store environment, product availability, and marketing strategies through interacting with retailers across China. Considering that e-cigarette retailers are predominately located in the most densely populated cities, the investigators will include approximately 1,080 e-cigarette retailers from 36 cities, including 4 municipalities directly under the Central Government, 27 provincial capital cities, and 5 cities specially designated in the state plan. Store addresses and contact information will be obtained through web scraping from the AutoNavi map (the most popular map app in China). The investigators plan to randomly sample 32 retailers in each city if the number allows, and cities with less than 32 retailers identified will all be included. To capture reality, retailers will not be informed during visit. The sampled ones within each city will be randomized into the intervention and control group, with a balance gender ratio of the simulated clients. These clients will be recruited from university students younger than 20 years old, who can easily be considered as minors (under 18) when purely judged by their appearance. Clients visiting retailers in the control group will dress in school uniforms and carry a school bag, while those in the intervention group will dress in professional attire with a business-style backpack for males or a leather bag for females. The clients will record retailer responses, including (1) inquiring about age verbally, (2) requesting identity cards for age verification, and (3) whether retailers still sell products even when identity cards are not presented. For each e-cigarette retailer, the nearest tobacco retailer identified through the AutoNavi Map will be used for comparison to document the differences in the behaviors between the two types of retailers. Additionally, communication and marketing strategies, e.g., mentioning available flavored products, dissuading clients not to purchase, are also collected.

ELIGIBILITY:
Inclusion Criteria:

* Retailers can be identified from the AutoNavi Map through keyword searches
* Retailers have reachable contact information
* Retailers are contacted and claim being open for business on a regular basis
* Include only one retailer if multiple ones have the same contact information

Exclusion Criteria:

* Retailers that are not located in main districts of the cities (usually old town and economically developed central areas)
* Perceived danger surrounding the retailers (e.g., remote alleys with no pedestrians at all)
* Closed when arriving
* Retailers that cannot be located based on map information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1089 (Actual)
Dates: Start 2023-07-29 (Actual); Primary Completion 2023-09-03 (Actual); Study Completion 2023-09-03 (Actual)

PRIMARY OUTCOMES:
Non-compliant sales | During visit (day 1)
  The simulated clients will report whether retailers sell e-cigarette products to possible minors even when identity cards are not presented for age verification.

SECONDARY OUTCOMES:
Inquiring about age | During visit (day 1)
  The simulated clients will report whether retailers inquire about their age verbally in stores.
Requesting identity cards | During visit (day 1)
  The simulated clients will report whether retailers request them to show identity cards for the purpose of age verification.

OTHER OUTCOMES:
Online contact | During visit (day 1)
  The simulated clients will report if they are able to add retailers as WeChat (the online most popular chat app in China) contacts.
Delivery service offered | During visit (day 1)
  The simulated clients will report if salespersons mention that products ordered online can be delivered to them.
Illegal flavored e-cigarette products available | During visit (day 1)
  The simulated clients will report if salespersons mention that flavored (non-national-standard) e-cigarette products are available in stores.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Wang, PhD, Principal Investigator — Peking University Health Science Center; Hai Fang, PhD, Principal Investigator — Peking University Health Science Center
Locations (1):
- 36 major metropolitan areas (Beijing included), Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Derived] Wang Y, Lv X, Laestadius LI, Guidry JPD, Mahmoudi E, Kong G, Chang J, Martin A, Yang M, Yan D, Si L, Bustamante AV, Fang H. E-Cigarette Sales to School-Uniformed Adolescents in China: A Randomized Clinical Trial. JAMA Netw Open. 2025 Oct 1;8(10):e2535623. doi: 10.1001/jamanetworkopen.2025.35623. PMID 41071555

DOCUMENTS (2):
  • Study Protocol (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT05962411/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT05962411/SAP_001.pdf